CLINICAL TRIAL: NCT04411667
Title: Randomized Open Label Study of Standard of Care Plus Intravenous Immunoglobulin (IVIG) Compared to Standard of Care Alone in the Treatment of COVID-19 Infection
Brief Title: Study of SOC Plus IVIG Compared to SOC Alone in the Treatment of COVID-19
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: George Sakoulas, MD (Other)
Collaborators: Octapharma (Industry)
Responsible Party: Sponsor-Investigator, George Sakoulas, MD, Infectious Disease Specialist, Sharp HealthCare
Organization: Sharp HealthCare (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID-IVIG; 2004902 (Other: Sharp HealthCare Institutional Review Board (SHC IRB))
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Results first posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Sars-CoV2
Keywords: Coronavirus; IVIG; COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Octagam; Immunoglobulins, Intravenous

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into one of two groups: Standard of Care plus IVIG or Standard of Care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (study drug+SOC) (Experimental): Standard of care plus IVIG (Octagam) 0.5g/kg IVPB actual body weight daily x 3 days, with premedication methylprednisolone 40 mg IV push x 1 30-50 minutes before each IVIG infusion. Initial infusion rate of IVIG (Octagam) will be of 0.6 mL/kg/hour, increasing to a maximum rate of 100ml/hr, if tolerated.
  Interventions: Drug: Octagam
- Group B (SOC) (No Intervention): Standard of Care

INTERVENTIONS:
Drug: Octagam — Standard of Care plus Octagam infusion for 3 days.
  Other Names: IVIG
  Arms: Group A (study drug+SOC)

SUMMARY:
The purpose of this research is to see if Intravenous Immunoglobulin (IVIG) can help reduce respiratory complications (respiratory failure and need for a ventilator) caused by coronavirus disease 2019 (COVID-19). The principal investigator has successfully utilized IVIG for patients infected with the influenza virus. The investigator wants to find out if IVIG is equally effective in COVID-19 infection patients, and if IVIG will give the immune system some help to clear the infection naturally.

DETAILED DESCRIPTION:
This is an investigator initiated, open label, multicenter, two arm, randomized study to compare the impact of adding IVIG to the Standard of Care (SOC) to the SOC without IVIG. Randomization will be 1:1. The goal of this study is to identify whether or not IVIG can halt the progression to respiratory failure requiring mechanical ventilation in subjects admitted to the hospital with confirmed COVID-19. The addition of IVIG to the standard of care treatment for these patients may be beneficial in abating acute lung injury in subjects with SARSCoV-2 induced hypoxia that results in organ injury.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 positive test result (including presumptive positive).
* Hospitalization
* Requiring ≥4 liters/min O2 nasal cannula to maintain oxygen saturation ≥ 92%, but not mechanically ventilated
* Age ≥18 years old.
* Access to a phone in the hospital room or an electronic device that is capable of receiving phone calls and/or video calls and/or e-mail.
* Able to read/write/speak English or Spanish fluently.
* Subjects must have the capacity to provide consent or an appropriate Legally Authorized Representative (LAR) to provide informed consent.

provide informed consent, and provide authorization of use and disclosure of personal health information.

* Negative pregnancy test for women of childbearing potential.

Exclusion Criteria:

* Severe allergy to any IVIG product formulation
* History of DVT, PE, thromboembolic stroke or other thrombotic events
* Hypersensitivity to corn. Octagam® contains maltose which is a sugar derived from corn.
* Uncontrolled hypertension (SBP>180 mm Hg or DBP>120mmHg)
* Active participant in another research treatment study
* Mechanically ventilated patient
* Code status is Do Not Resuscitate or Do Not Intubate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Sakoulas, MD, Principal Investigator — Sharp HealthCare
Locations (2):
- United States (2):
  - Sharp Grossmont Hospital, La Mesa, California
  - Sharp Memorial Hospital, San Diego, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A (Study Drug+SOC) | Group B (SOC)
Started | 17 | 17
Completed | 16 | 17
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Study Drug+SOC) | Group B (SOC) | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Full Range); unit: years] | 54 [27 to 69] | 54 [19 to 80] | 54 [19 to 80]
Age, Continuous [Median (Full Range); unit: years] | 59 [27 to 69] | 51 [19 to 80] | 56 [19 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 15 | 28
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 32.5 [20.8 to 49.6] | 34.9 [22.7 to 51.9] | 33.6 [20.8 to 51.9]
Comorbidities [Count of Participants; unit: Participants]
  Diabetes mellitus | 6 | 6 | 12
  Hypertension | 4 | 7 | 11
  Chronic kidney disease | 0 | 1 | 1
  Coronary artery disease | 1 | 1 | 2
  Congestive heart failure | 1 | 1 | 2
  Asthma/chronic obstructive pulmonary disease | 2 | 2 | 4
  Current smoker | 1 | 1 | 2
  Former smoker | 2 | 1 | 3
  Immunocompromised | 1 | 0 | 1
Comorbidities Continued (HbA1c) [Mean (Full Range); unit: % glycosylated hemoglobin] | 10.1 [9 to 12.9] | 6.4 [4.8 to 7.3] | 8.1 [4.8 to 12.9]
Other Coronavirus Disease 2019 Therapies [Count of Participants; unit: Participants]
  Remdesivir | 8 | 9 | 17
  Convalescent plasma | 2 | 3 | 5
  Glucocorticoids | 16 | 10 | 26

OUTCOME MEASURES:

1. Primary Outcome: Mechanical Ventilation
Description: Number of subjects requiring mechanical ventilation due to respiratory failure
Time Frame: from date of patient admission to date of patient discharge or date of death, whichever came first, assessed up to 45 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Study Drug+SOC) | Group B (SOC)
Number analyzed (Participants) | 16 | 17
Participants | 2 | 7

2. Secondary Outcome: Oxygen Therapy
Description: Number of days requiring oxygen therapy
Time Frame: as for outcome 1
Population: This data was not collected although it was originally intended to be an outcome measure
Arm/Group | Group A (Study Drug+SOC) | Group B (SOC)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Length of Stay
Description: Number of days in hospital
Time Frame: from date of patient admission to date of patient discharge or date of death, whichever came first, assessed up to 60 days
Measure: Median (Full Range); unit: days
Arm/Group | Group A (Study Drug+SOC) | Group B (SOC)
Number analyzed (Participants) | 16 | 17
days | 12 [6 to 29] | 17 [4 to 60]

ADVERSE EVENTS:
Time Frame: from date of patient enrollment to date of patient discharge or date of death, whichever came first, assessed up to 45 days
Arm/Group | Group A (Study Drug+SOC) | Group B (SOC)
All-Cause Mortality (participants affected / at risk) | 1/16 | 3/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 7/16 | 8/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Study Drug+SOC) (N=16) | Group B (SOC) (N=17)
Elevated D-Dimer (General disorders) | 2 (2) | 2 (2)
Acute Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Elevated Liver Function Tests (General disorders) | 3 (3) | 0 (0)
Hyperglycemia (General disorders) | 3 (3) | 2 (2)
Thrombocytosis (General disorders) | 1 (1) | 1 (1)
Anemia (General disorders) | 0 (0) | 3 (3)
Leukocytosis (General disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
* Study limited to two hospitals in one US city. Resulted in a homogenous population of younger Hispanic/Latino patients.
* Study was not blinded.
* Methylprednisolone was used as a pre-medication for each dose of IVIG which may have confounded the results.
* Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT04411667/Prot_SAP_000.pdf